CLINICAL TRIAL: NCT03100929
Title: The Efficiency in Nuchal Cord Detection in Sonographic Evaluation as Performed by an Unexperienced First Year Resident With Minimal Training.
Brief Title: Nuchal Cord Detection in Sonographic Evaluation by a First Year Resident.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, ROY LAUTERBACH MD, Principal Investigator, Rambam Health Care Campus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0405-16-RMB
Record Dates: First submitted 2017-03-29; First posted 2017-04-04 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Fetal Cord Entanglement
MeSH Terms: conditions — Nuchal Cord | interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Elective cesarean section (Experimental): Any patient undergoing elective cesarean section. Ultrasound
  Interventions: Diagnostic Test: Ultrasound

INTERVENTIONS:
Diagnostic Test: Ultrasound — Pre-operational ultrasound for the detection of fetal heart rate, fetal presentation and presence of nuchal cord.

SUMMARY:
The investigators aim to prove that minimal sonographic training for nuchal cord detection in an unexperienced first year medical resident is more than enough to detect the phenomenon. Patients undergoing elective cesarean section will undergo a routine ultrasound (that is performed to detect the fetal heart rate and the fetal presentation) during which the resident will attempt to detect nuchal cord. The resident will then attend the patient's surgery to verify the findings.

DETAILED DESCRIPTION:
Patients undergoing elective cesarean section will undergo a routine ultrasound examination during which fetal heart rate, fetal presentation and nuchal cord presence will be documented. During surgery, after the fetus is delivered, presence or lack of nuchal cord will be documented.

The aim of the study is to show that minimal sonographic training may assist even an unexperienced sonographist in detection of such a subtle yet important phenomenon.

The study will be performed utilizing the newest resident in the OBGYN department.

ELIGIBILITY:
Inclusion Criteria:

* Any woman undergoing elective cesarean section.

Exclusion Criteria:

* None.

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female-term pregnancy.
Enrollment: 100 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Detection rate for nuchal cord. | up to 6 hours from admission for elective surgery.
  Detection of nuchal cord in a pre-op ultrasound and verification of the sonographic findings during surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Roy Lauterbach, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam health care campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No